CLINICAL TRIAL: NCT06002594
Title: The Effects of Two Different Nasal Irrigation Techniques on Physiological Parameters, Crying Duration, and Feeding in Relieving Nasal Congestion in Infants
Brief Title: Examination of the Effectiveness of Nasal Irrigation Techniques in Infants With Nasal Congestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nevin Avsar, nurse, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sislietfal-SBF-NAG-01
Record Dates: First submitted 2023-08-06; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Upper Respiratory Tract Infection; Nasal Congestion and Inflammations
Keywords: infants; nasal irrigation; nasal lavage; feeding
MeSH Terms: conditions — Respiratory Tract Infections; Nasal Obstruction; Inflammation

STUDY DESIGN:
Intervention Model Description: two groups were randomly selected and received two different treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group low-volume irrigation (Experimental): Nasal irrigation was performed using low-volume saline solution
  Interventions: Other: group low-volume irrigation
- group high-volume irrigation (Experimental): Nasal irrigation was performed using high-volume saline solution
  Interventions: Other: group high-volume irrigation

INTERVENTIONS:
Other: group low-volume irrigation — Before the procedure, infants' physiological parameters were measured using the Nellcor Bedside SpO2 Patient Monitoring System. The procedure duration and crying duration were recorded using the stopwatch on a Samsung Galaxy A50 phone. Nasal irrigation was performed using 4 ml of 0.9% sodium chloride(NaCl) solution. Physiological parameters were measured immediately after the procedure and five minutes later. Subsequently, breastfeeding was initiated for the baby. Physiological parameters during breastfeeding were measured, and parental satisfaction levels were evaluated. Then, the frequency of procedure repetitions was recorded.
  Arms: group low-volume irrigation
Other: group high-volume irrigation — Before the procedure, infants' physiological parameters were measured using the Nellcor Bedside SpO2 Patient Monitoring System. The procedure duration and crying duration were recorded using the stopwatch on a Samsung Galaxy A50 phone. Nasal irrigation was performed using 20 ml of 0.9% NaCl solution. Physiological parameters were measured immediately after the procedure and five minutes later. Subsequently, breastfeeding was initiated for the baby. Physiological parameters during breastfeeding were measured, and parental satisfaction levels were evaluated. Then, the frequency of procedure repetitions was recorded.
  Arms: group high-volume irrigation

SUMMARY:
The research investigates the effects of high-volume and low-volume nasal irrigation techniques applied to relieve nasal congestion in infants with nasal congestion due to upper respiratory tract infections. The study examines the physiological parameters of infants who undergo nasal irrigation, crying duration, frequency of the procedure, and the baby's feeding patterns.

DETAILED DESCRIPTION:
This study aims to investigate the effects of two different nasal irrigation techniques applied to relieve nasal congestion on infants' physiological parameters, crying duration, feeding habits, and the frequency of the procedure repetitions.

A randomized controlled experimental study was conducted with 80 infants aged 1-12 months who presented at the pediatric emergency clinic with nasal congestion due to upper respiratory tract infection. In the study, the 1st group of infants received low-volume saline solution, while the 2nd group received high-volume saline solution for nasal irrigation. Physiological parameters were measured before the procedure, immediately after the procedure, and 5 minutes after the procedure. Procedure duration and baby's crying duration were recorded. Subsequently, breastfeeding was initiated for the infants, and their physiological parameters were measured again during breastfeeding. Parental satisfaction levels with the procedure were also assessed. Finally, the frequency of the procedure repetitions was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with Upper Respiratory Tract Infection and recommended nasal cleaning with saline solution by a physician,
* Infants whose parents provided consent for their participation in the research,
* Term-born infants aged 1 month to 12 months,
* Breastfed infants,
* Infants without chronic illnesses,
* Conscious infants,

Exclusion Criteria:

* Infants with congenital anomalies affecting the respiratory system (such as choanal atresia, etc.),
* Infants with allergic rhinitis,
* Infants who used antibiotics or corticosteroids before hospital admission,
* Infants with growth retardation, were excluded from the study.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
The Effect of Low-Volume and High-Volume Nasal Irrigation Techniques on Infant's Physiological Parameters | 3 months
  Prior to low and high-volume nasal irrigation procedures, infants' average peripheral oxygen saturation (SpO2), average heart rate per minute, and average respiratory rate per minute will be measured immediately before the procedure, immediately after the procedure, and five minutes after the procedure. The aim is to examine the effect of irrigation on physiological parameters.

SECONDARY OUTCOMES:
The Effect of Nasal Irrigation Procedure on Procedure Duration, Infant Crying Duration, and Procedure Repetition Frequency | 3 months
  Since the irrigation procedure can be distressing for the infant, two stopwatches were initiated to measure the duration of crying associated with the procedure. One was started just before the nasal irrigation procedure, and the other when the infant began crying. The first stopwatch was stopped after the procedure, while the second stopwatch was stopped when the infant's crying ceased. For infants with persistent post-irrigation nasal congestion, the procedure was repeated at 15-minute intervals, and the number of procedure repetitions was recorded.

OTHER OUTCOMES:
The Impact of Nasal Irrigation Techniques on Infant Feeding | 3 months
  After the nasal irrigation procedures, breastfeeding was initiated. During breastfeeding, average peripheral oxygen saturation (SpO2), average heart rate per minute, and average respiratory rate per minute were recorded. Following breastfeeding, mothers were asked to assess their current breastfeeding performance compared to the baby's performance before the procedure, and their satisfaction level with the procedure was recorded by inquiring about their level of contentment.

CONTACTS AND LOCATIONS:
Overall Officials: Nevin AVŞAR GÖK, Principal Investigator — University of Health Sciences Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- University of Health Sciences Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Sarıyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No